CLINICAL TRIAL: NCT04854863
Title: Respiratory Muscle Function After Hospitalisation for COVID-19 -Pathophysiological Model on Severity, Determinants and Clinical Consequences of Respiratory Muscle Strength Impairment in Patients Who Had Been Hospitalised for COVID-19-
Brief Title: Respiratory Muscles After Hospitalisation for COVID-19
Acronym: REMAP-COVID-19
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Jens Spießhöfer, Jens Spiesshoefer, MD, PhD Candidate, Group Head Respiratory Physiology, RWTH Aachen University
Other Study IDs: CTCA 20-515
Record Dates: First submitted 2021-04-15; First posted 2021-04-22 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Covid19; Diaphragm Injury
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples obtained based on venous puncture
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Comprehensive assessment of respiratory muscle function. — Comprehensive assessment of respiratory muscle function to the point of its invasive assessment with recordings of twitch transdiaphragmatic pressure in response to magnetic phrenic nerve stimulation and stimulation of the lower thoracic nerve roots.

SUMMARY:
Fatigue and exercise intolerance after survived COVID-19-infection might be related to weakness of the respiratory muscles especially following invasive mechanical ventilation in the Intensive Care Unit.

The aim of the project is to measure respiratory muscle function and strength in our respiratory physiology laboratory (Respiratory Physiology Laboratory, Department of Pneumology and Intensive Care Medicine, Head: Professor Michael Dreher) in patients who survived a severe COVID-19-infection (25 with a severe course requiring mechanical ventilation in the intensive care unit, 25 with a moderate-severe course requiring administration of supplemental oxygen only, respectively).

Based on this data the aim is to develop a model which determines the severity, pathophysiology and clinical consequences of respiratory muscle dysfunction in patients who had been hospitalised for COVID-19.

This will potentially prove the importance of a dedicated pulmonologic rehabilitation with respiratory muscle strength training in patients who had been hospitalised for COVID-19.

DETAILED DESCRIPTION:
The aim of the present project is to comprehensively measure respiratory muscle function and strength in patients who survived a hospitalisation for a severe COVID-19-infection (25 with a severe course requiring mechanical ventilation in the intensive care unit, 25 with a moderate-severe course requiring administration of supplemental oxygen only, respectively).

We intend to recruit 50 patients during their regular follow up appointments (12 months and 24 months after their discharge from the hospital) in our pulmonology outpatient-clinic. Patients fulfilling the criterions of inclusion and exclusion will be included.

Patients will undergo a series of measurements on one day in our respiratory physiology laboratory (Respiratory Physiology Laboratory, Department of Pneumology and Intensive Care Medicine, Head: Professor Michael Dreher). Patients will be asked to complete a questionnaire, followed by some examinations comprising spirometry by bodyplethysmography, exercise endurance, capillary blood gas analyses, measurement of maximum inspiratory and expiratory mouth pressures, dynamometric measurement of arm and leg strength, diaphragm ultrasound, magnetic stimulation of the phrenic and lower thoracic nerves with invasive recording of twitch transdiaphragmatic pressure and markers of systemic inflammation based on in depth analyses of blood samples that will be obtained.

Based on this data the aim is to develop a model which determines the severity, pathophysiology and clinical consequences of respiratory muscle dysfunction in patients who had been hospitalised for COVID-19.

This will potentially prove the importance of a dedicated pulmonologic rehabilitation with respiratory muscle strength training in patients who had been hospitalised for COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* 50 patients with survived COVID-19-infection (25 with a severe course requiring mechanical ventilation in the intensive care unit, 25 with a moderate-severe course requiring administration of supplemental oxygen only, respectively)
* Patients aged at least 18 years, who are mentally and physically able to consent and participate into the study

Exclusion Criteria:

* Diagnosis of another disease, which causes a permanent increase in carbon dioxide level in the blood (chronic hypercapnia) or a permanent combined lung weakness (particularly a neuromuscular disease)
* Body-mass-index (BMI) >40
* Expected absence of active participation of the patient in study-related measurements
* Alcohol or drug abuse
* Metal implant in the body that is not MRI compatible (NON MRI compatible pacemaker, implantable defibrillator, cervical implants, e.g. brain pacemakers etc.)
* Slipped disc
* Epilepsy
* Bound to a wheel chair
* Patients who are mentally and physically unable to consent and participate into the study
* Patients in an interdependence or with an employment contract with the principal investigator, Co-PI or his deputy.
* Emergency hospital stay in the last 4 weeks preceding the day of the measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The aim of the present project is to comprehensively measure respiratory muscle function and strength in patients who survived a hospitalisation for a severe COVID-19-infection (25 with a severe course requiring mechanical ventilation in the intensive care unit, 25 with a moderate-severe course requiring administration of supplemental oxygen only, respectively)
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Twitch transdiaphragmatic pressure in response to supramaximal magnetic stimulation of the phrenic nerve roots | 2 years
  Recording of twitch transdiaphragmatic pressure (Unit: Pressure in cmH2O)
Respiratory mouth pressures | 2 years
  Measurement of respiratory (inspiratory and expiratory) mouth pressures (Unit: Pressure in cmH2O)

SECONDARY OUTCOMES:
Diaphragm ultrasound | 2 years
  Comprehensive evaluation of diaphragm excursion (amplitude during tidal breathing, sniff maneuver and maximal inspiration in cm, corresponding velocity in cm/sec, respectively) and thickening on ultrasound (thickness at functional residual capacity, at total lung capactiy in cm), Markers of Diaphragm excursion and thickening will be combined to classify diaphragm function as normal, mildly, moderately or severly impaired.
Exercise intolerance | 2 years
  Comprehensive evaluation of symptoms (breathlesness based on NYHA class, on a visual scale ranging from 1-10, respectively) and exercise capacity (6 minute walking distance). These measurements will be combined to classifiy patients as presenting with exercise intolerance or no exercise intolerance.
Analyses of markers of systemic inflammation (interleukin levels in ng/ml, TNF alpha in ng/ml, CRP in mg/L; immune phenotyping of inflammatory cells, most importantly whilte blood cell subtypes in %) | 2 years
  Analyses of markers of systemic inflammation based on blood samples taken. These measurements will be combined to classify patients as having increased or normal levels of systemic inflammation.
Lung function | 2 years
  Comprehensive assessment of lung function by bodyplethysmography (most importantly forced vital capacity, forced expiratory volume after 1 second, intrathoracic gas volume, residual volume) and capillary blood gas analysis (most importantly pO2 in mmHG and pCO2 in mmHG). These measurements will be combined to classify patients as showing normal, restrictive, obstructive lung function impairment, as being hypoxic, hypercapnic, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dreher, Professor, Study Director — RWTH Aachen University; Jens Spiesshoefer, MD, Principal Investigator — RWTH Aachen University; Janina Friedrich, MD, Study Chair — RWTH Aachen University
Locations (1):
- Jens Spiesshoefer, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Daher A, Balfanz P, Aetou M, Hartmann B, Muller-Wieland D, Muller T, Marx N, Dreher M, Cornelissen CG. Clinical course of COVID-19 patients needing supplemental oxygen outside the intensive care unit. Sci Rep. 2021 Jan 26;11(1):2256. doi: 10.1038/s41598-021-81444-9. PMID 33500431
- [Background] Daher A, Balfanz P, Cornelissen C, Muller A, Bergs I, Marx N, Muller-Wieland D, Hartmann B, Dreher M, Muller T. Follow up of patients with severe coronavirus disease 2019 (COVID-19): Pulmonary and extrapulmonary disease sequelae. Respir Med. 2020 Nov-Dec;174:106197. doi: 10.1016/j.rmed.2020.106197. Epub 2020 Oct 20. PMID 33120193
- [Background] Balfanz P, Hartmann B, Muller-Wieland D, Kleines M, Hackl D, Kossack N, Kersten A, Cornelissen C, Muller T, Daher A, Stohr R, Bickenbach J, Marx G, Marx N, Dreher M. Early risk markers for severe clinical course and fatal outcome in German patients with COVID-19. PLoS One. 2021 Jan 29;16(1):e0246182. doi: 10.1371/journal.pone.0246182. eCollection 2021. PMID 33513168
- [Background] Spiesshoefer J, Henke C, Herkenrath S, Brix T, Randerath W, Young P, Boentert M. Transdiapragmatic pressure and contractile properties of the diaphragm following magnetic stimulation. Respir Physiol Neurobiol. 2019 Aug;266:47-53. doi: 10.1016/j.resp.2019.04.011. Epub 2019 Apr 25. PMID 31029769
- [Background] Spiesshoefer J, Henke C, Herkenrath S, Randerath W, Brix T, Young P, Boentert M. Assessment of Central Drive to the Diaphragm by Twitch Interpolation: Normal Values, Theoretical Considerations, and Future Directions. Respiration. 2019;98(4):283-293. doi: 10.1159/000500726. Epub 2019 Jul 26. PMID 31352459
- [Background] Spiesshoefer J, Herkenrath S, Henke C, Langenbruch L, Schneppe M, Randerath W, Young P, Brix T, Boentert M. Evaluation of Respiratory Muscle Strength and Diaphragm Ultrasound: Normative Values, Theoretical Considerations, and Practical Recommendations. Respiration. 2020;99(5):369-381. doi: 10.1159/000506016. Epub 2020 May 12. PMID 32396905
- [Derived] Spiesshoefer J, Regmi B, Senol M, Jorn B, Gorol O, Elfeturi M, Walterspacher S, Giannoni A, Kahles F, Gloeckl R, Dreher M. Potential Diaphragm Muscle Weakness-related Dyspnea Persists 2 Years after COVID-19 and Could Be Improved by Inspiratory Muscle Training: Results of an Observational and an Interventional Clinical Trial. Am J Respir Crit Care Med. 2024 Sep 1;210(5):618-628. doi: 10.1164/rccm.202309-1572OC. PMID 38763165
- [Derived] Regmi B, Friedrich J, Jorn B, Senol M, Giannoni A, Boentert M, Daher A, Dreher M, Spiesshoefer J. Diaphragm Muscle Weakness Might Explain Exertional Dyspnea 15 Months after Hospitalization for COVID-19. Am J Respir Crit Care Med. 2023 Apr 15;207(8):1012-1021. doi: 10.1164/rccm.202206-1243OC. PMID 36596223
- [Derived] Spiesshoefer J, Friedrich J, Regmi B, Geppert J, Jorn B, Kersten A, Giannoni A, Boentert M, Marx G, Marx N, Daher A, Dreher M. Diaphragm dysfunction as a potential determinant of dyspnea on exertion in patients 1 year after COVID-19-related ARDS. Respir Res. 2022 Jul 15;23(1):187. doi: 10.1186/s12931-022-02100-y. PMID 35841032